CLINICAL TRIAL: NCT00315939
Title: Improving Metabolic Control and Reducing Hypoglycemic Risk in Type 1 Diabetes Mellitus With Biological and Behavioral Feedback
Brief Title: Improving Control and Reducing the Risk of Hypoglycemic Episodes in Type 1 Diabetes
Acronym: BPK002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boris Kovatchev, PhD (Other)
Responsible Party: Sponsor-Investigator, Boris Kovatchev, PhD, Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 12126
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; hypoglycemic episodes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A Order: SMBG, IBMF-1, IBMF-2 (Experimental): Group A performed routine self-monitored blood glucose (SMBG) alone (level 1), followed sequentially by Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1) level 2 and Integrated Biobehavioral Monitoring & Feedback - 2 (IBMF-2) level 3. Each level continued for 3 months.
  Interventions: Device: Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1); Device: Integrated Biobehavioral Monitoring & Feedback - 2 (IBMF-2)
- Group B Order: IBMF-1, IBMF-2, SMBG (Experimental): Group B began with Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1) level 2, followed by level 3, Integrated Biobehavioral Monitoring & Feedback - 2 (IBMF-2) and then level 1 (SMBG only). Each level continued for 3 months.
  Interventions: Device: Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1); Device: Integrated Biobehavioral Monitoring & Feedback - 2 (IBMF-2)

INTERVENTIONS:
Device: Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1) — Integrated Biobehavioral Monitoring & Feedback-1 (IBMF-1): a hand-held computer (HHC) was given to the subjects, programmed to estimate HbA1c, risk for hypoglycemia (Low BG Index), and glucose variability (Average Daily Risk Range) using previously published algorithms. The subjects were asked to carry the HHC and enter all their self-monitored blood glucose (SMBG) readings. The estimates of HbA1c were updated weekly, and the estimates of risk for hypoglycemia and glucose variability were updated at each SMBG entry. Detailed instructions were provided on the meaning of these different types of glucose feedback; the study staff was available to answer any questions.
Device: Integrated Biobehavioral Monitoring & Feedback - 2 (IBMF-2) — Integrated Biobehavioral Monitoring & Feedback-2 (IMBF-2) retains IMBF-1, but the HHC asked subjects to provide symptom ratings when blood glucose (BG) was low and at an equal number of matching euglycemic readings. From these data, the HHC estimated a set of potentially significant symptoms of hypoglycemia for each individual, using an iterative algorithm following a previously published symptom significance estimation procedure. The patient manual for the HHC program is provided in supplementary data of published manuscript.

SUMMARY:
The purpose of this study is to test two newly developed computer programs, Integrated Biobehavioral Monitoring and Feedback (IBMF) IBMF-1 and IBMF-2. The computer programs are considered experimental. Both computer programs are being tested to see if they are useful in helping people with type 1 diabetes avoid low blood sugar episodes.

DETAILED DESCRIPTION:
Subjects were randomized into group A or group B matched by gender, age, and baseline HbA1c. Group A began with routine self-monitored blood glucose (SMBG) alone (level 1), followed sequentially by IBMF-1 (level 2) and IBMF-2 (level 3). Group B began with level 2, followed by level 3 and then level 1.

Each level continued for 3 months and proceeded as follows: level 1 was routine SMBG. Subjects were given LifeScan OneTouch UltraSmart meters (LifeScan Inc., Milpitas, CA) and free strips, and asked to perform SMBG four to five times per day. No additional instructions about the timing of SMBG or the interpretation of the data were given. No changes to treatment were recommended. At each visit, the subject was only asked about any health concerns or any new medications or change in insulin. This information was recorded but not used for feedback. Thus, level 1 should be regarded as a control condition, which was different from routine SMBG only because subjects were enrolled in a study and given free test strips.

IBMF-1 (level 2) retained level 1, but an HHC (hand-held computer) was given to the subjects, programmed to estimate HbA1c, risk for hypoglycemia (Low BG Index, LBGI), and glucose variability (Average Daily Risk Range, ADRR) using previously published algorithms. The subjects were asked to carry the HHC and enter all their glucose readings when per- forming SMBG. The estimates of HbA1c were updated weekly, and the estimates of risk for hypoglycemia and glucose variability were updated at each SMBG entry. Detailed instructions were provided on the meaning of these different types of glucose feedback; the study staff was available to answer any questions.

IBMF-2 (level 3) retained level 2, but the HHC asked subjects to provide symptom ratings when BG (blood glucose) was low and at an equal number of matching euglycemic readings. From these data, the HHC estimated a set of potentially significant symptoms of hypoglycemia for each individual, using an iterative algorithm following a previously published symptom significance estimation procedure. The patient manual for the HHC program is provided in supplementary data of published manuscript.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have type 1 diabetes as defined by the American Diabetes Association or by the judgment of the physician
* Willing to participate for up to one year
* Perform routine blood glucose checks 3-4 times a day
* Complete monthly diaries of the occurrence of severe and moderate hypoglycemic episodes
* Have 6 hemoglobin A1c (HgbA1c) drawn
* Have a mixed meal tolerance test to assess for residual pancreatic insulin secretion

Exclusion Criteria:

* Age < 18 years
* Currently abusing alcohol or drugs
* Severe depression or psychosis
* Significant mental impairment
* Inability to use a glucometer and a hand held computer
* Pregnant or desire to achieve pregnancy within the following year (females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Kovatchev, Ph.D., Principal Investigator — University of Virginia, Department of Psychiatric Medicine, Behavioral Medicine Research
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Kovatchev BP, Mendosa P, Anderson S, Hawley JS, Ritterband LM, Gonder-Frederick L. Effect of automated bio-behavioral feedback on the control of type 1 diabetes. Diabetes Care. 2011 Feb;34(2):302-7. doi: 10.2337/dc10-1366. Epub 2011 Jan 7. PMID 21216860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 120 adults with type 1 diabetes were recruited through regional advertising. Inclusion criteria were age ≥18 years, type 1 diabetes defined by the American Diabetes Association criteria or physician judgment, and willingness to participate in the study for up to 12 months performing finger sticks four to five times per day.
Groups:
- Experimental: Group A Order: SMBG, IBMF-1, IBMF-2: Self-monitored blood glucose (SMBG) alone (level 1), followed sequentially by Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1) level 2 and IBMF-2, level 3. IBMF-1 (level 2) retained level 1, but an HHC (hand-held computer) was given to the subjects, programmed to estimate HbA1c, risk for hypoglycemia, and glucose variability. The subjects were asked to carry the HHC and enter all their glucose readings when performing SMBG. The estimates of HbA1c were updated weekly, and the estimates of risk for hypoglycemia and glucose variability were updated at each SMBG entry. IBMF-2 (level 3) retained level 2, but the HHC asked subjects to provide symptom ratings when BG (blood glucose) was low and at an equal number of matching euglycemic readings. From these data, the HHC estimated a set of potentially significant symptoms of hypoglycemia for each individual, using an iterative algorithm following a previously published symptom significance estimation procedure.
- Experimental: Group B Order: IBMF-1, IBMF-2, SMBG: Integrated Biobehavioral Monitoring & Feedback - 1 (IBMF-1) level 2 followed by IBMF-2, level 3 and then SMBG only. IBMF-1 (level 2) retained level 1, but an HHC (hand-held computer) was given to the subjects, programmed to estimate HbA1c, risk for hypoglycemia, and glucose variability. The subjects were asked to carry the HHC and enter all their glucose readings when performing SMBG. The estimates of HbA1c were updated weekly, and the estimates of risk for hypoglycemia and glucose variability were updated at each SMBG entry. IBMF-2 (level 3) retained level 2, but the HHC asked subjects to provide symptom ratings when BG (blood glucose) was low and at an equal number of matching euglycemic readings. From these data, the HHC estimated a set of potentially significant symptoms of hypoglycemia for each individual, using an iterative algorithm following a previously published symptom significance estimation procedure.
Period: Admission 1 (3 Months)
Arm/Group | Experimental: Group A Order: SMBG, IBMF-1, IBMF-2 | Experimental: Group B Order: IBMF-1, IBMF-2, SMBG
Started | 59 | 61
Completed | 56 | 55
Not Completed | 3 | 6
Period: Admission 2 (3 Months)
Arm/Group | Experimental: Group A Order: SMBG, IBMF-1, IBMF-2 | Experimental: Group B Order: IBMF-1, IBMF-2, SMBG
Started | 56 | 55
Completed | 52 | 51
Not Completed | 4 | 4
Period: Admission 3 (3 Months)
Arm/Group | Experimental: Group A Order: SMBG, IBMF-1, IBMF-2 | Experimental: Group B Order: IBMF-1, IBMF-2, SMBG
Started | 52 | 51
Completed | 48 | 49
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Group A Order: SMBG, IBMF-1, IBMF-2: Group A will perform routine SMBG alone (level 1), followed sequentially by levels 2 and 3. Each level continued for 3 months.
- Experimental: Group B Order: IBMF-1, IBMF-2, SMBG: Group B will begin with level 2, followed by level 3 and then level 1. Each level will continue for 3 months.
- Total: Total of all reporting groups
Arm/Group | Experimental: Group A Order: SMBG, IBMF-1, IBMF-2 | Experimental: Group B Order: IBMF-1, IBMF-2, SMBG | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.65 (14.84) | 37.61 (13.78) | 39.15 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Time Frame: 1 year (each level lasted 3 months)
Population: All 120 participants were analyzed; data for subjects who dropped out during the study were handled according to the intention-to-treat principle, using "dropout" as a factor and adjusting significance levels accordingly. Below data for the 97 participants who completed the 1-year protocol are shown.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Groups:
- Experimental Groups A and B: Group A: SMBG alone (level 1), followed sequentially by levels 2 and 3. Group B: Level 2, followed by level 3 and then level 1.
  Each level continued for 3 months.
  IBMF-1 (level 2) retained level 1, but an HHC (hand-held computer) was given to the subjects, programmed to estimate HbA1c, risk for hypoglycemia, and glucose variability. The subjects were asked to carry the HHC and enter all their glucose readings when performing SMBG. The estimates of HbA1c were updated weekly, and the estimates of risk for hypoglycemia and glucose variability were updated at each SMBG entry.
  IBMF-2 (level 3) retained level 2, but the HHC asked subjects to provide symptom ratings when BG (blood glucose) was low and at an equal number of matching euglycemic readings. From these data, the HHC estimated a set of potentially significant symptoms of hypoglycemia for each individual, using an iterative algorithm following a previously published symptom significance estimation procedure.
Arm/Group | Experimental Groups A and B
Number analyzed (Participants) | 97
percentage of glycated hemoglobin
  Baseline | 7.99 (1.48)
  Post-Level 1 | 7.69 (1.30)
  Post-Level 2 | 7.69 (1.33)
  Post-Level 3 | 7.58 (1.08)
Statistical Analysis 1: Comparison: Experimental Groups A and B; Test type: Superiority or Other; p = 0.001, ANOVA

2. Primary Outcome: Frequency of Severe Hypoglycemia
Description: Severe hypoglycemia (SH) was defined to subjects as "blood glucose so low that you could not treat yourself because you were stuporous or unconscious."
Time Frame: 1 year (each level lasted 3 months)
Population: as for outcome 1
Measure: Number; unit: episodes/month/person
Arm/Group | Experimental Groups A and B
Number analyzed (Participants) | 97
episodes/month/person
  SH Baseline | 0.09
  SH Post-Level 1 | 0.21
  SH Post-Level 2 | 0.15
  SH Post-Level 3 | 0.02

ADVERSE EVENTS:
Time Frame: January 2006 - December 2009
Groups:
- IBMF-1: IBMF-1 will use the OneTouch® UltraSmart® glucometer (LifeScan, Milpitas, CA) to collect routine SMBG data and the subject transfers the blood glucose (BG) value into a hand-held computer (HHC) for processing. As the subject checks BG on a daily basis, the IBMF-1 software calculates an estimate of HbA1c, acute risk for hypoglycemia and chronic risk for hypoglycemia. This information will be presented back to the subject. Specifically, (i) alarms for immediate action if BG<50 mg/dL is registered; (ii) a running HbA1c estimate (71); (iii) a warning to be more careful and measure BG more frequently over the next 24 hours if elevated acute risk for hypoglycemia is found, and (iv) an indication of the subject's chronic risk for hypoglycemia in one of 4 categories (minimal, low, moderate, and high). At moderate and high risk the subject will be prompted to consider altering his/her behavior. HbA1c and chronic risk change slowly (2-3 weeks), while acute risk can change daily.
- IBMF-2: IBMF-2 retains level 2, but the HHC asks subjects to provide symptom ratings when BG (blood glucose) is low and at an equal number of matching euglycemic readings. From these data, the HHC estimates a set of potentially significant symptoms of hypoglycemia for each individual, using an iterative algorithm following a previously published symptom significance estimation procedure.
Arm/Group | IBMF-1 | IBMF-2
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/107
Other Adverse Events (participants affected / at risk) | 0/117 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No